CLINICAL TRIAL: NCT06326320
Title: The Effects of Combined Serratus Anterior Plane Block on Postoperative Acute Pain After Minimally Invasive Cardiac Surgery
Brief Title: Combined SAPB in MICS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Nilgün Zengin, Principal İnvestigator, Ankara City Hospital Bilkent
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E.Kurul-E2-24-6175
Record Dates: First submitted 2024-03-17; First posted 2024-03-22 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Serratus Anterior Plane Block; Acute Pain; Postoperative Analgesia; Minimal Invasive Cardiac Surgery
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Combined serratus anterior plane block (Other): Following the visualization of the anatomical structures, the nerve block needle will be advanced via the in-plane technique beneath the serratus anterior muscles until the interfascial space was reached. After hydrodissection with 2 ml normal saline, 20 ml 0.25% bupivacaine will be injected into the area. Then, with the same needle, will be returned 1-2 cm from the deep serratus anterior area to superficial serratus anterior area above the serratus anterior muscle and will be injected 2 ml normal saline for hydrodissection. Finally 20ml of 0.25% bupivacaine will be injected for superficial serratus anterior block into the interfacial area.
  Interventions: Procedure: Combined SAPB

INTERVENTIONS:
Procedure: Combined SAPB — Combined Deep and Superficial Serratus Anterior Plane Block will be performed unilaterally, under US guidance, before the surgical operation, after the induction of anesthesia, when the patient is placed in the supine position. 40 ml of 0.25% bupivacaine will be used in applications.

SUMMARY:
Minimally invasive cardiac surgery (MICS) has begun to be performed frequently in recent years. Compared to sternotomy, MISC reduces the risk of mediastinitis, leaves a more aesthetic scar, facilitates postoperative rehabilitation, and shortens the hospital stay. MICS requires a thoracic incision in the right 4th or 5th intercostal space. This incision causes intense and long-lasting pain in the postoperative period. Pain is exacerbated by breathing movements, coughing, and respiratory physiotherapy.

Postoperative analgesia is a critical risk factor for the development of pulmonary and cardiovascular complications in any type of cardiothoracic surgery. If patients with high pain levels cannot breathe effectively, it may lead to atelectasis, cardiac ischemia, and arrhythmias. This prolongs the time it takes for patients to be discharged and increases the frequency of postoperative pulmonary complications and postoperative morbidity.

In addition to intravenous medications, various neuraxial and peripheral nerve blocks can be used in cardiac surgery. In recent years, thoracic epidural analgesia has been avoided due to the use of intraoperative high-dose heparin. As an alternative, peripheral nerve blocks have recently gained popularity. SAPB is one of them. SAPB can be applied in three ways. While deep SAPB (DSAPB) is applied under the serratus anterior muscle, superficial SAPB (SSAPB) is applied above the serratus anterior muscle. Combined SAPB (CSAPB) is applied both below and above the serratus anterior muscle. These blocks can be performed with a single injection anywhere between the second and seventh ribs on the lateral chest wall.

In this study, the analgesic effects of ultrasound-guided CSAPB application in patients undergoing MICS will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 80 years old
* American Society of Anesthesiologists (ASA) physical status I-II-III
* BMI 18 to 40 kg/m2
* Elective Minimally Invasive Cardiac Surgery (MICS)

Exclusion Criteria:

* Patient refusing the procedure
* Emergency surgery
* History of chronic opioid or analgesic used

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-06-10 (Actual); Study Completion 2025-06-25 (Actual)

PRIMARY OUTCOMES:
Pain Scores | 0th hour the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 0th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 2nd hour the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 2nd-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 4th hour the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 4th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 8th hour the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 8th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).
Pain Scores | 12th hour the extubation
  After the extubation, pain will be assessed for the sternum and the drain area at the 12th-hour rest and while coughing using the visual analog scale on a scale from 0 (no pain) to 10 (worst pain).

SECONDARY OUTCOMES:
Remifentanyl Consumption | intraoperative period
  Remifentanyl consumption for intraoperative period will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara City Hospital, Çankaya, Ankara, Turkey (Türkiye)